CLINICAL TRIAL: NCT06564233
Title: A Randomized Controlled Trial of an Avatar-based Supportive Care Intervention for Patients Undergoing Outpatient Stem Cell Transplantation
Brief Title: Supportive Care Intervention for Outpatient Stem Cell Transplant Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friendi.fi Corporation (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); care.coach corporation (Industry)
Responsible Party: Principal Investigator, Victor Wang, Co-founder, President, Friendi.fi Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DFCI 24-183
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cancer
Keywords: health coaching; conversational relational agents
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- care.coach Avatar™ (Experimental): care.coach Avatar™ with usual supportive care. The avatar program includes companionship, HCT educational modules, relaxation and mindfulness exercises, simple (seated) physical exercises, nightly check ins, and symptom self-management as needed.
  Interventions: Behavioral: care.coach Avatar™
- Usual Supportive Care (No Intervention): Traditional supportive care comprising of a binder with HCT educational materials and regular meetings with a transplant nurse.

INTERVENTIONS:
Behavioral: care.coach Avatar™ — care.coach Avatar™ ("avatar") is a conversational relational agent that serves as a virtual companion and appears on a tablet device as an animated pet avatar. Each avatar is supervised by a 24x7 remote team of trained human staff whose abilities are augmented by artificial intelligence (AI) and software-driven health coaching and clinical protocols for consistency, automation, and scale. This unique human-in-the-loop design enables safe, empathic, natural conversations that form the basis for trusting relations and lasting behavior change. In addition to being a companion, the avatar educates patients about their condition, helps manage symptoms, and reinforces other healthy habits. Independent studies have demonstrated improved outcomes at a reduced cost of care. A pilot study demonstrated the feasibility of care.coach Avatar™ as a psychosocial support and health coach in hospitalized HCT patients. More research is needed to assess efficacy and applications in other HCT settings.
  Arms: care.coach Avatar™

SUMMARY:
The overall goal of this study is to assess the efficacy of the care.coach Avatar™ in improving anxiety and quality of life for patients undergoing outpatient transplant. After care.coach Avatar™ content and scheduling ("digital intervention" or "program") has been optimized for outpatient allogeneic hematopoietic stem cell transplantation (HCT), a randomized controlled trial (RCT) will be conducted of the digital versus usual supportive care program for outpatient HCT recipients. Potential improvements in anxiety and quality of life will be evaluated, with the intent of increasing comfortability with outpatient transplant and expanding the population of eligible patients willing to receive their transplants in an outpatient setting.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HCT) is the delivery of multipotent donor-derived stem cells to a recipient patient. It typically involves a lengthy inpatient hospitalization (median 25.8 days). With improving availability of health services, prophylactic medications, and lower infection risk and transfusion requirements, outpatient HCT is becoming more prevalent for patients receiving reduced intensity conditioning (RIC). However, even for outpatient HCT, patients are hospitalized for a median of 8 days. Most symptoms from HCT are concentrated in the first 30-days after the transplant, and these must be better addressed to optimize benefits from outpatient HCT. For patients undergoing HCT, incidence of psychological consequences is higher than in other cancer health states; potential psychological symptoms include stress, anxiety, anger, depression, insomnia, and loneliness. Non-pharmacological approaches for improving quality of life (QOL) and reducing distress among HCT patients include psychoeducational, exercise, and mindfulness interventions. Although post-HCT changes in lifestyle are challenging, the Health Belief Model and Prochaska's Transtheoretical model of change posit that patients preparing for HCT day 0 (notated as D0), when they receive the stem cell infusion, would be highly motivated to learn about psychosocial supports and activities given their readiness for change and taking action. This presents an ideal timeframe for studying a psychosocial health coaching intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Seen for outpatient RIC HCT (prior to D0, generally D-6).

Exclusion Criteria:

* Deemed by clinical staff or research assistant (RA) to be unable to converse with an avatar, due to: severe, uncorrectable hearing or vision impairment; severe speech impairment that precludes understanding by staff (or by the avatar).
* Not fluent in English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HADS-A | Baseline, Day 20 (D+20) post-transplant
  Hospital Anxiety and Depression Scale (HADS) - Anxiety subscale

SECONDARY OUTCOMES:
FACT-BMT | Baseline, Day 20 (D+20) post-transplant
  Functional Assessment of Cancer Therapy - Bone Marrow Transplantation
HADS-A | Baseline, Day 90 (D+90) post-transplant
  Hospital Anxiety and Depression Scale (HADS) - Anxiety subscale
FACT-BMT | Baseline, Day 90 (D+90) post-transplant
  Functional Assessment of Cancer Therapy - Bone Marrow Transplantation

OTHER OUTCOMES:
Conversions | Day 20 (D+20) post-transplant, Day 90 (D+90) post-transplant
  Conversion from Outpatient to Inpatient Transplant
HADS-D | Baseline, Day 20 (D+20) post-transplant, Day 90 (D+90) post-transplant
  Hospital Anxiety and Depression Scale (HADS) - Depression subscale

CONTACTS AND LOCATIONS:
Overall Officials: Victor Wang, MS, Principal Investigator — Friendi.fi Corporation; Chantal M Kerssens, PhD, Study Director — Friendi.fi Corporation
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT06564233/ICF_000.pdf